CLINICAL TRIAL: NCT04211974
Title: Genomic Landscape of Intramedullary Astrocytoma
Acronym: GIMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Fengzeng Jian, director of neurospine department, Xuanwu hospital, Xuanwu Hospital, Beijing
Other Study IDs: Xuanwu-IMA
Record Dates: First submitted 2019-12-24; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Spinal Cord Astrocytoma
Keywords: spinal cord astrocytoma; whole-exome sequencing;
MeSH Terms: interventions — Exome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor resected and matched blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: whole-exome sequencing — Fresh frozen or formalin-fixed, paraffin-embedded samples were obtained from patients following resection along with matching peripheral blood samples.
  whole-exome sequencing will be performed to identify mutations in tumor tissue and matching blood

SUMMARY:
intramedullary astrocytoma is a rare and devastating spinal cord glioma. while the management of intracranial astrocytoma includes gross total resection, radiotherapy and chemotherapy, spinal cord astrocytoma is very difficult to be totally removed due to its infiltrative nature and unclear plane of dissection; Moreover, the use radiotherapy and chemotherapy for spinal cord astrocytoma is controversial. Therefore, the treatment for spinal cord astrocytoma is very limited as compared to its intracranial counterpart. Inadequate understanding of spinal cord astrocytoma mainly contribute to limited treatment, while the molecular profiling of intracranial astrocytoma is relatively well understood. Hence, we performed whole-exome sequencing of intramedullary astrocytoma aiming to identify the pathophysiological mechanisms underlying spinal cord astrocytoma

DETAILED DESCRIPTION:
Intramedullary tumor only account for 2-4% of central nervous tumor. Of which, ependymoma and astrocytoma represent the most common intramedullary tumor. Although intramedullary astrocytoma is rare, it can cause significant mortality and morbidity. Different from its intracranial counterpart which can receive gross total resection and standard adjuvant treatment, intramedullary astrocytoma always cannot be removed completed due to its infiltrative nature and, additionally, radiotherapy and chemotherapy is controversial. Therefore, the treatment for this tumor is very limited. While the genetic profiling of intracranial astrocytoma is relatively well understood and standard treatment strategy has been developed, genetic alteration of intramedullary astrocytoma is less well understood. Identification of the molecular profiling can lead to well understanding of the pathophysiological mechanisms underlying intramedullary astrocytoma and more effective therapeutic strategy in future. Hence, we performed this study aiming to investigate the genetic profiling of intramedullary. All patients with intramedullary astrocytoma underwent surgery in our institution will be enrolled. Tumor tissue and matching blood will be obtained after the surgery. Whole-exome sequencing was performed on DNA extracted from these specimens. Moreover, demographic information, progress-free survival and overall survival will be evaluated in 3 year of follow-up after the initial diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* patients that histologically diagnosed as primary spinal cord astrocytoma

Exclusion Criteria:

* patients with spinal cord tumors rather than astrocytoma
* metastatic astrocytoma
* tumor sample can not be obtained

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who was histologically diagnosed as primary spinal cord astrocytoma or was suspected of primary spinal cord astrocytoma will be enrolled. But patiens who was suspected of primary spinal cord astrocytoma preoperatively but was confirmed as tumor rather than astrocytoma postoperatively via histology will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
molecular profiling results | 1 month after the surgery
  mutation identified via whole-exome sequencing will be recored.

SECONDARY OUTCOMES:
overall survival | 3 years after the diagnosis
  overall survival of patients with spinal cord astrocytoma will be recorded;defined as the duration from the date of diagnosis to the date of final follow-up or death
progression free survival | 3 years after the diagnosis
  progression free survival of patients with spinal cord astrocytoma will be recorded;was defined as the duration from the date of diagnosis to the date of tumor progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Fengzeng Jian, Study Director — Xuanwu Hospital, Capitial Medical University
Locations (1):
- Xuanwu Hospital, China International Neuroscience Institute, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ogunlade J, Wiginton JG 4th, Elia C, Odell T, Rao SC. Primary Spinal Astrocytomas: A Literature Review. Cureus. 2019 Jul 26;11(7):e5247. doi: 10.7759/cureus.5247. PMID 31565645
- [Background] Nabors LB, Portnow J, Ammirati M, Baehring J, Brem H, Butowski N, Fenstermaker RA, Forsyth P, Hattangadi-Gluth J, Holdhoff M, Howard S, Junck L, Kaley T, Kumthekar P, Loeffler JS, Moots PL, Mrugala MM, Nagpal S, Pandey M, Parney I, Peters K, Puduvalli VK, Ragsdale J, Rockhill J, Rogers L, Rusthoven C, Shonka N, Shrieve DC, Sills AK, Swinnen LJ, Tsien C, Weiss S, Wen PY, Willmarth N, Bergman MA, Engh A. NCCN Guidelines Insights: Central Nervous System Cancers, Version 1.2017. J Natl Compr Canc Netw. 2017 Nov;15(11):1331-1345. doi: 10.6004/jnccn.2017.0166. PMID 29118226
- [Background] Guss ZD, Moningi S, Jallo GI, Cohen KJ, Wharam MD, Terezakis SA. Management of pediatric spinal cord astrocytomas: outcomes with adjuvant radiation. Int J Radiat Oncol Biol Phys. 2013 Apr 1;85(5):1307-11. doi: 10.1016/j.ijrobp.2012.11.022. Epub 2013 Feb 20. PMID 23433793
- [Background] Kim WH, Yoon SH, Kim CY, Kim KJ, Lee MM, Choe G, Kim IA, Kim JH, Kim YJ, Kim HJ. Temozolomide for malignant primary spinal cord glioma: an experience of six cases and a literature review. J Neurooncol. 2011 Jan;101(2):247-54. doi: 10.1007/s11060-010-0249-y. Epub 2010 Jun 5. PMID 20526650
- [Background] Chi JH, Cachola K, Parsa AT. Genetics and molecular biology of intramedullary spinal cord tumors. Neurosurg Clin N Am. 2006 Jan;17(1):1-5. doi: 10.1016/j.nec.2005.10.002. No abstract available. PMID 16448901
- [Background] McGirt MJ, Goldstein IM, Chaichana KL, Tobias ME, Kothbauer KF, Jallo GI. Extent of surgical resection of malignant astrocytomas of the spinal cord: outcome analysis of 35 patients. Neurosurgery. 2008 Jul;63(1):55-60; discussion 60-1. doi: 10.1227/01.NEU.0000335070.37943.09. PMID 18728568
- [Result] Milano MT, Johnson MD, Sul J, Mohile NA, Korones DN, Okunieff P, Walter KA. Primary spinal cord glioma: a Surveillance, Epidemiology, and End Results database study. J Neurooncol. 2010 May;98(1):83-92. doi: 10.1007/s11060-009-0054-7. Epub 2009 Nov 7. PMID 19898743
- [Result] Adams H, Avendano J, Raza SM, Gokaslan ZL, Jallo GI, Quinones-Hinojosa A. Prognostic factors and survival in primary malignant astrocytomas of the spinal cord: a population-based analysis from 1973 to 2007. Spine (Phila Pa 1976). 2012 May 20;37(12):E727-35. doi: 10.1097/BRS.0b013e31824584c0. PMID 22609727
- [Result] Liu A, Sankey EW, Bettegowda C, Burger PC, Jallo GI, Groves ML. Poor prognosis despite aggressive treatment in adults with intramedullary spinal cord glioblastoma. J Clin Neurosci. 2015 Oct;22(10):1628-31. doi: 10.1016/j.jocn.2015.05.008. Epub 2015 Jun 30. PMID 26142051
- [Result] Karsy M, Guan J, Sivakumar W, Neil JA, Schmidt MH, Mahan MA. The genetic basis of intradural spinal tumors and its impact on clinical treatment. Neurosurg Focus. 2015 Aug;39(2):E3. doi: 10.3171/2015.5.FOCUS15143. PMID 26235020
- [Result] Fakhreddine MH, Mahajan A, Penas-Prado M, Weinberg J, McCutcheon IE, Puduvalli V, Brown PD. Treatment, prognostic factors, and outcomes in spinal cord astrocytomas. Neuro Oncol. 2013 Apr;15(4):406-12. doi: 10.1093/neuonc/nos309. Epub 2013 Jan 14. PMID 23322747
- [Result] Moinuddin FM, Alvi MA, Kerezoudis P, Wahood W, Meyer J, Lachance DH, Bydon M. Variation in management of spinal gliobastoma multiforme: results from a national cancer registry. J Neurooncol. 2019 Jan;141(2):441-447. doi: 10.1007/s11060-018-03054-2. Epub 2018 Nov 20. PMID 30460627
- [Result] Shows J, Marshall C, Perry A, Kleinschmidt-DeMasters BK. Genetics of Glioblastomas in Rare Anatomical Locations: Spinal Cord and Optic Nerve. Brain Pathol. 2016 Jan;26(1):120-3. doi: 10.1111/bpa.12327. No abstract available. PMID 26443345
- [Result] Zhang M, Iyer RR, Azad TD, Wang Q, Garzon-Muvdi T, Wang J, Liu A, Burger P, Eberhart C, Rodriguez FJ, Sciubba DM, Wolinsky JP, Gokaslan Z, Groves ML, Jallo GI, Bettegowda C. Genomic Landscape of Intramedullary Spinal Cord Gliomas. Sci Rep. 2019 Dec 10;9(1):18722. doi: 10.1038/s41598-019-54286-9. PMID 31822682
- [Result] Shankar GM, Lelic N, Gill CM, Thorner AR, Van Hummelen P, Wisoff JH, Loeffler JS, Brastianos PK, Shin JH, Borges LF, Butler WE, Zagzag D, Brody RI, Duhaime AC, Taylor MD, Hawkins CE, Louis DN, Cahill DP, Curry WT, Meyerson M. BRAF alteration status and the histone H3F3A gene K27M mutation segregate spinal cord astrocytoma histology. Acta Neuropathol. 2016 Jan;131(1):147-50. doi: 10.1007/s00401-015-1492-2. No abstract available. PMID 26487540